CLINICAL TRIAL: NCT05537220
Title: NAC Attack, A Phase III, Multicenter, Randomized, Parallel, Double Masked, Placebo-Controlled Study Evaluating the Efficacy and Safety of Oral N-Acetylcysteine in Patients With Retinitis Pigmentosa
Brief Title: Oral N-acetylcysteine for Retinitis Pigmentosa
Acronym: NAC Attack
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Duke University (Other); Emory University (Other); Massachusetts Eye and Ear Infirmary (Other); Mayo Clinic (Other); Medical College of Wisconsin (Other); Retina Foundation of the Southwest (Other); Stanford University (Other); University of California, Davis (Other); University of Florida (Other); University of Iowa (Other); University of Miami (Other); University of Michigan (Other); University of Minnesota (Other); University of Oklahoma (Other); University of Southern California (Other); University of Utah (Other); University of Washington (Other); University of Wisconsin, Madison (Other); Vanderbilt University (Other); Vitreo Retinal Associates, PA (Unknown); University of Houston (Other); Medical University of Graz (Other); McGill University (Other); Universität Tübingen (Other); Radboud University Medical Center (Other); University of Amsterdam (Other); University Hospital, Basel, Switzerland (Other); University College London Hospitals (Other); Northwestern University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00337490; 2022-003023-17 (EudraCT Number); 1UG1EY033293 (NIH); 2022-501438-46-00 (Other: Clinical Trials Application)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa
Keywords: N-acetylcysteine; Ellipsoid zone; Macular sensitivity; Best corrected visual acuity; Ellipsoid zone width; Ellipsoid zone area; Oxidative damage; Usher Syndrome; Antioxidants
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 483 participants will be enrolled and randomized at approximately 30 clinical sites in the Americas and Europe. Patients will be eligible if both eyes have an RP phenotype consisting of severe loss of rod function (night blindness) followed by progressive constriction of visual fields with best-corrected visual acuity (BCVA) of 20/60 or better. Gradable ellipsoid zone (EZ) width on the horizontal fovea spectral domain-optical coherence tomography (SD-OCT) scan must be < 8000 µm and ≥ 1500 µm. Eligible patients will be randomized 2:1 to NAC 1800 mg bid versus placebo. The primary efficacy objective is to determine if the progressive loss in EZ width measured as the cumulative loss of EZ (calculated as the area above the curve) between baseline and month (M) 45 is significantly less in eyes of participants taking NAC 1800 mg bid compared with that in eyes of participants taking placebo. The safety objective is to evaluate the long-term safety and tolerability of oral NAC for 45 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - N-acetylcysteine (Experimental): This is the intervention group. Patients in this group will be receiving 1800 mg of N-acetylcysteine in the form of 3 effervescent 600 mg tablets dissolved in water twice a day for 45 months.
  Interventions: Drug: N-acetylcysteine
- Group 2 - Placebo (Placebo Comparator): Patients in the placebo group will receive identical effervescent tablets lacking active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — After randomization, participants will be given about 10-months supply of study drug (intervention), with instructions to take 3 effervescent tablets in water twice a day. They will return to the clinic at M4.5 for evaluation and then at M9, M18, M27, M36, M40.5 and M45. At each in-clinic visit, drug reconciliation will occur. At each visit at Baseline, M9, M18, M27, M36, that is, every 9 months, participants will be given another 10-month supply of study drug.
  Arms: Group 1 - N-acetylcysteine
Drug: Placebo — After randomization, participants will be given about 10-months supply of placebo, with instructions to take 3 effervescent tablets in water twice a day. They will return to the clinic at M4.5 for evaluation and then at M9, M18, M27, M36, M40.5 and M45. At each in-clinic visit, efficacy and safety assessments will be done and drug reconciliation will occur. At baseline, M9, M18, M27, and M36 participants will be given another 10-month supply of placebo.
  Arms: Group 2 - Placebo

SUMMARY:
Retinitis pigmentosa (RP) is an inherited retinal degeneration caused by one of several mistakes in the genetic code. Such mistakes are called mutations. The mutations cause degeneration of rod photoreceptors which are responsible for vision in dim illumination resulting in night blindness. After rod photoreceptors are eliminated, gradual degeneration of cone photoreceptors occurs resulting in gradual constriction of side vision that eventually causes tunnel vision. Oxidative stress contributes to cone degeneration. N-acetylcysteine (NAC) reduces oxidative stress and in animal models of RP it slowed cone degeneration. In a phase I clinical trial in patients with RP, NAC taken by month for 6 months caused some small improvements in two different vision tests suggesting that long-term administration of NAC might slow cone degeneration in RP. NAC Attack is a clinical trial being conducted at many institutions in the US, Canada, and Europe designed to determine if taking NAC for several years provides benefit in patients with RP.

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP) is a disease in which one of several different mutations differentially causes degeneration of rod photoreceptors while sparing cone photoreceptors. The loss of rod photoreceptors results in poor vision in dim illumination (night blindness), but does not affect most activities of daily life including reading or driving. However, after most rod photoreceptors are eliminated, cone photoreceptors begin to die, resulting in gradual constriction of visual fields which over time causes visual disability.

Rods outnumber cones by a ratio of 95:5 and therefore after mutation-induced degeneration of rods, the majority of cells in the outer retina have been eliminated, markedly reducing oxygen utilization. However, oxygen supply is unchanged resulting in a large excess of tissue oxygen surrounding cones. This results in progressive oxidative damage that contributes to slowly progressive degeneration of cone photoreceptors. N-acetylcysteine (NAC) is a strong antioxidant that is approved for acetaminophen overdose. Orally administered NAC in a mouse model of RP reduced oxidative damage to cones and promoted maintenance of function and survival of cones. In a phase I clinical trial in patients with RP, oral administration of NAC for 6 months was well-tolerated and resulted in a small but statistically significant improvement in visual acuity and light sensitivity in the retina. This suggests that long-term administration of NAC may promote survival and maintenance of function of cones. NAC Attack is a phase III, multicenter, randomized, placebo controlled trial that will determine if oral NAC provides benefit and is safe in patients with RP.

ELIGIBILITY:
Inclusion Criteria:

General

* Ability and willingness to provide informed consent
* Age ≥ 18 and ≤65 years at time of signing Informed Consent Form
* Ability and willingness to comply with the study protocol and to participate in all study visits and assessments in the investigator's judgement
* For candidates of childbearing potential: willingness to use a method of contraception
* Agreement not to take supplements other than vitamin A

Ocular Inclusion Criteria

* Both eyes must exhibit the RP phenotype with evidence of loss of night vision, gradual constriction of visual fields, and maintenance of visual acuity;
* In addition, an eye must meet the following criteria to be included in the study:
* Gradable EZ on a horizontal SD-OCT scan through the fovea center with width ≤ 8000 µm and ≥1500 µm and with well-defined truncation at both the nasal and temporal sides;
* BCVA ≥ ETDRS letter score of 61 (20/60 Snellen equivalent);
* Sufficiently clear ocular media and adequate pupillary dilation to allow good quality images sufficient for analysis and grading by central reading center.

Exclusion Criteria:

General Exclusion Criteria

* Active cancer within the past 12 months, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer with Gleason score ≤ 6 and stable prostate specific antigen for > 12 months
* Renal failure requiring renal transplant, hemodialysis, peritoneal dialysis, or anticipated to require hemodialysis or peritoneal dialysis during the study
* Liver disease, cystic fibrosis, asthma, or chronic obstructive pulmonary disease (COPD), history of thrombocytopenia not due to a reversible cause or other blood dyscrasia
* Uncontrolled blood pressure (defined as systolic > 180 and/or diastolic > 100 mmHg while at rest) at screening. If a patient's initial measurement exceeds these values, a second reading may be taken 30 or more minutes later. If the patient's blood pressure must be controlled by antihypertensive medication, the patient may become eligible if medication is taken continuously for at least 30 days.
* History of other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion that oral NAC may be contraindicated or that follow up may be jeopardized
* Cerebrovascular accident or myocardial infarction within 6 months of screening
* Participation in an investigational study that involves treatment with any drug or device within 6 months of screening
* Three relatives already enrolled in study
* Pregnant, breast feeding, or intending to become pregnant during the study treatment period. Women of childbearing potential who have not had tubal ligation must have a urine pregnancy test at screening.
* Known history of allergy to NAC
* Having taken NAC in any form in the past 4 months
* Phenylketonuria
* Fructose intolerance
* Glucose-galactose malabsorption
* Sucrase-isomaltase insufficiency
* Abnormal laboratory value including the value of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin being greater than 1.5 x the upper limit of normal
* Any major abnormal findings on blood chemistry, hematology, and renal function lab tests that in the opinion of the Site Investigator and/or the Study Chair makes the candidate not suitable to participate in the trial
* HIV or hepatitis B infection

Ocular Exclusion Criteria

* Evidence of cone-rod dystrophy or pattern dystrophy including focal areas of atrophy or pigmentary changes in the central macula
* Cystoid spaces involving the fovea substantially reducing vision
* Glaucoma or other optic nerve disease causing visual field loss or reduced visual acuity
* Intra ocular pressure >27 mm Hg from two measurements. If a patient's initial measurement exceeds 27 mm Hg, a second reading must be taken.
* Any retinal disease other than RP causing reduction in visual field or visual acuity
* Any prior macular laser photocoagulation
* Intraocular surgery within 3 months prior to screening
* High myopia with spherical equivalent refractive error > 8 diopters. If an eye has had cataract surgery or refractive surgery, a pre-operative refractive error spherical equivalent > 8 diopters is an exclusion
* Any concurrent ocular condition that might affect interpretation of results
* History of uveitis in either eye

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Progressive change of ellipsoid zone (EZ) width | Baseline and 45 months
  The EZ is a hyperreflective band seen on SD-OCT scans that corresponds to photoreceptors with intact inner and outer segments. In RP patients at the stage of those participating in this trial, the EZ consists primarily of remaining cones with intact inner and outer segments. The EZ width is the length of the EZ on a horizontal SD-OCT scan through the fovea and provides a quantitative measure of surviving cones. The primary outcome measure is the progressive change (loss) in EZ width measured as the cumulative loss of EZ (calculated as the area above the curve) between baseline and month (M) 45.

SECONDARY OUTCOMES:
Change in mean macular sensitivity measured by microperimetry (MP) | Baseline and 45 months
  The macula is the functional center of the retina. Macular sensitivity is a measure of the sensitivity to light assessed at focal points within the macula. It is measured by microperimetry (MP), a test in which light stimuli of many different intensities are presented at multiple loci in the macula and the response or lack of response to those stimuli are recorded. Sensitivity is determined by the weakest light stimulus that is detected at a locus. The mean macular sensitivity is the average of the sensitivity measurements at the test loci and provides a quantitative assessment of macula function.
Change in best-corrected visual acuity | Baseline and 45 months
  Visual acuity is the vision mediated by the fovea (the center of the macula) that is used for fine visual tasks including reading and driving. In order to measure the best-corrected visual acuity (BCVA), it is necessary to eliminate all refractive error with lenses to optimally focus images on the fovea. This is done using a standardized protocol established in the Early Treatment Diabetic Retinopathy Study (ETDRS); it measures the number of letters read at 4 meters on a standardized chart under standardized lighting conditions. Since the fovea is made up of cones, BCVA is a measure of cone function.

OTHER OUTCOMES:
Cumulative change of EZ area assessed as the area above curve (AAC) | Baseline and 45 months
  EZ area is determined by measuring EZ width of multiple horizontal SD-OCT scans ranging from the superior to the inferior part of the macula. A line drawn connecting contiguous points where the EZ ends provides a 3-dimensional map of the region where there are photoreceptors with intact inner and outer segments.
Change in mean macular sensitivity measured by MP | Baseline, 4.5 months, 9 months, 18 months, 27 months, 36 months, 40.5 months
  To assess whether compared to placebo, NAC promotes maintenance of macular function, it is necessary to compare the two study groups over a long period of time. It is useful to determine how differences in mean macular sensitivity between the two groups evolve over time and therefore an exploratory outcome is change in mean macular sensitivity between baseline and each time point at which it is measured throughout the study.
Change in BCVA | Baseline, 4.5 months, 9 months, 18 months, 27 months, 36 months, 40.5 months
  To assess whether compared to placebo, NAC promotes maintenance of BCVA, it is necessary to compare the two study groups over a long period of time. It is useful to determine how differences in BCVA between the two groups evolve over time and therefore an exploratory outcome is change in BCVA between baseline and each time point at which it is measured throughout the study.
Change in cone spacing measured by adaptive optics-scanning laser ophthalmoscopy (AOSLO) | Baseline, 9 months, 27 months, 45 months
  AOSLO provides unique ability to monitor cones at single cell resolution over time. As cone degeneration occurs, there is reduction in cone density even in areas where EZ is intact and therefore assessment of cone spacing by AOSLO provides a more sensitive assessment of cone health than SD-OCT derived EZ measurements. This will provide an anatomical assessment of the efficacy of NAC and will help evaluate the feasibility of using AOSLO-derived outcome measures in future interventional studies in RP.
Change in cone regularity measured by AOSLO | Baseline, 9 months, 27 months, 45 months
  AOSLO provides unique ability to monitor cones at single cell resolution over time. As cone degeneration occurs, there is reduction in cone density even in areas where EZ is intact and therefore assessment of cone regularity by AOSLO provides a more sensitive assessment of cone health than SD-OCT derived EZ measurements. This will provide an anatomical assessment of the efficacy of NAC and will help evaluate the feasibility of using AOSLO-derived outcome measures in future interventional studies in RP.
Change in cone reflectivity measured by AOSLO | Baseline, 9 months, 27 months, 45 months
  Measurements of EZ width and EZ area provide assessments of remaining cones with intact inner and outer segments, but do not have the resolution to assess individual cone structure and density. AOSLO provides unique ability to monitor cones at single cell resolution over time. As cone degeneration occurs, there is reduction in cone density even in areas where EZ is intact and therefore assessment of cone reflectivity by AOSLO provides a more sensitive assessment of cone health than SD-OCT derived EZ measurements. This will provide an anatomical assessment of the efficacy of NAC and will help evaluate the feasibility of using AOSLO-derived outcome measures in future interventional studies in RP.
Proportion of eyes with ≥ 5 loci change (improvement) from baseline by ≥ 6 decibels (dB) | Baseline, 4.5 months, 9 months, 18 months, 27 months, 36 months, 40.5 months, 45 months
  Mean macular sensitivity provides a global assessment of macular function. In addition to this global assessment, It is also useful to assess changes at individual loci which is afforded by MP. A change of 6 dB at a locus is unlikely to be due to chance, because it is well above test-retest variability and it is approximately 2 times the standard deviation of the locus level sensitivity changes that were seen in RP patients treated with NAC for 6 months. A useful assessment of whether or not NAC provides benefit in the macula of patients with RP is to determine if compared to eyes of participants treated with placebo, a greater proportion of eyes of participants treated with NAC have 5 or more loci with change (improvement) from baseline ≥ 6 dB at M4.5, M9, M18, M27, M36, M40.5, and M45.
Proportion of eyes with ≥ 5 loci change (decrease) from baseline by ≥ 6 decibels (dB) | Baseline, 4.5 months, 9 months, 18 months, 27 months, 36 months, 40.5 months, 45 months
  In addition to determining if more macular loci show improvement ≥ 6 dB in eyes of RP patients treated with NAC versus eyes of RP patients treated with placebo, it is important to determine if fewer macular loci show a change (decrease) ≥ 6 dB in eyes of RP patients treated with NAC versus eyes of RP patients treated with placebo.
Change in patient reported outcome assessed using NEI-VFQ 25 | Baseline, 27 months, 45 months
  It is useful to obtain the perspective of patients regarding the impact of treatment on their activities of daily life and quality of life. This is provided by the National Eye Institute Visual Function Questionnaire 25 (VFQ-25), a short form of the National Eye Institute Visual Function Questionnaire (NEI-VFQ), a self reported 51 item questionnaire. It is scored from 0 to 100 that is meant to be a measure of the subject's visual ability. A higher score signifies good visual ability and a lower score signifies poor visual ability that is negatively impacting quality of life.
Safety of oral NAC as assessed by adverse events | 45 months
  Oral NAC has a good safety profile but this study will use a higher dose of NAC and a longer treatment period in a different patient population than any prior study. It is important to assess safety of long term administration of NAC 1800 mg bid in patients with RP. This will be assessed by determining the incidence of ocular and non-ocular adverse events (AEs) in participants treated with NAC versus those treated with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Study Chair — Johns Hopkins University; Xiangrong Kong, Study Director — Johns Hopkins University
Locations (31):
- United States (24):
  - University of California - Davis, Department of Ophthalmology & Vision Science, Davis, California
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - University of California - San Francisco, Department of Ophthalmology, San Francisco, California
  - Stanford University, Byers Eye Institute, Stanford, California
  - Vitreo Retinal Associates, Gainesville, Florida
  - University of Florida - Jacksonville, UF Health Jacksonville, Jacksonville, Florida
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Emory Eye Center, Atlanta, Georgia
  - University Of Illinois At Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Iowa, Carver College of Medicine, Iowa City, Iowa
  - Wilmer Eye Institute- Johns Hopkins University, Baltimore, Maryland
  - Harvard University, Mass. Eye and Ear, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - University of Minnesota, Department of Ophthalmology and Visual Neurosciences, Minneapolis, Minnesota
  - Mayo Clinic, Department of Ophthalmology, Rochester, Minnesota
  - University of Oklahoma, Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Vanderbilt University, Vanderbilt Eye Institute, Nashville, Tennessee
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Utah, Moran Eye Center, Salt Lake City, Utah
  - University of Washington, Department of Ophthalmology, Seattle, Washington
  - University of Wisconsin - Madison, McPherson Eye Research Institute, Madison, Wisconsin
  - Medical College of Wisconsin, The Eye Institute, Milwaukee, Wisconsin
- Medical University of Graz, Department of Ophthalmology, Graz, Styria, Austria
- McGill University, The Research Institute of the McGill University Health Center, Montreal, Quebec, Canada
- University of Tübingen, Department für Augenheilkunde, Tübingen, Baden-Wurttemberg, Germany
- Netherlands (2):
  - Radboud University, Radboud University Medical Centre, Nijmegen, Gelderland
  - University of Amsterdam, Amsterdam Medical Center, Amsterdam, Northern Holland
- Universitätsspital Basel, Eye Clinic, Basel, Switzerland
- University College London, Moorfields Eye Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accord with the NIH guidelines, a summary, de-identified NAC Attack data set will be made available through submission of the dataset to a government or other health research database. The investigators will share individual-participant level data (IPD) together with their associated data dictionaries. The rights and privacy of people who participated in the Study will be protected at all times by stripping all identifiers including study identification numbers that could lead to disclosing the identity of individual research participants from the data. This commitment to privacy-protected data sharing will be incorporated in all levels of data sharing activities. In addition, redacted clinical study reports, retinal images, and other summary reports may be provided to researchers upon approval of their requests by the study leadership. The requesting researchers will be required to sign a data use agreement before given access to study reports or images.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be made available 1 year after publication of the primary findings of the study, in a de-identified format.
  For how long will we share the data?
Access Criteria: The study data sharing will follow the NIH's Data Sharing Policy published in the NIH Guide on February 26, 2003.
URL: https://sharing.nih.gov/data-management-and-sharing-policy/about-data-management-and-sharing-policy/data-management-and-sharing-policy-overview

REFERENCES:
- [Background] Bunker CH, Berson EL, Bromley WC, Hayes RP, Roderick TH. Prevalence of retinitis pigmentosa in Maine. Am J Ophthalmol. 1984 Mar;97(3):357-65. doi: 10.1016/0002-9394(84)90636-6. PMID 6702974
- [Background] Haim M. Epidemiology of retinitis pigmentosa in Denmark. Acta Ophthalmol Scand Suppl. 2002;(233):1-34. doi: 10.1046/j.1395-3907.2002.00001.x. PMID 11921605
- [Background] Rivolta C, Sharon D, DeAngelis MM, Dryja TP. Retinitis pigmentosa and allied diseases: numerous diseases, genes, and inheritance patterns. Hum Mol Genet. 2002 May 15;11(10):1219-27. doi: 10.1093/hmg/11.10.1219. PMID 12015282
- [Background] Boughman JA, Vernon M, Shaver KA. Usher syndrome: definition and estimate of prevalence from two high-risk populations. J Chronic Dis. 1983;36(8):595-603. doi: 10.1016/0021-9681(83)90147-9. PMID 6885960
- [Background] Athanasiou D, Aguila M, Bellingham J, Li W, McCulley C, Reeves PJ, Cheetham ME. The molecular and cellular basis of rhodopsin retinitis pigmentosa reveals potential strategies for therapy. Prog Retin Eye Res. 2018 Jan;62:1-23. doi: 10.1016/j.preteyeres.2017.10.002. Epub 2017 Oct 16. PMID 29042326
- [Background] Cao SS, Kaufman RJ. Unfolded protein response. Curr Biol. 2012 Aug 21;22(16):R622-6. doi: 10.1016/j.cub.2012.07.004. No abstract available. PMID 22917505
- [Background] Bowes C, Li T, Danciger M, Baxter LC, Applebury ML, Farber DB. Retinal degeneration in the rd mouse is caused by a defect in the beta subunit of rod cGMP-phosphodiesterase. Nature. 1990 Oct 18;347(6294):677-80. doi: 10.1038/347677a0. PMID 1977087
- [Background] Chang B, Hawes NL, Pardue MT, German AM, Hurd RE, Davisson MT, Nusinowitz S, Rengarajan K, Boyd AP, Sidney SS, Phillips MJ, Stewart RE, Chaudhury R, Nickerson JM, Heckenlively JR, Boatright JH. Two mouse retinal degenerations caused by missense mutations in the beta-subunit of rod cGMP phosphodiesterase gene. Vision Res. 2007 Mar;47(5):624-33. doi: 10.1016/j.visres.2006.11.020. Epub 2007 Jan 30. PMID 17267005
- [Background] McLaughlin ME, Sandberg MA, Berson EL, Dryja TP. Recessive mutations in the gene encoding the beta-subunit of rod phosphodiesterase in patients with retinitis pigmentosa. Nat Genet. 1993 Jun;4(2):130-4. doi: 10.1038/ng0693-130. PMID 8394174
- [Background] Farber DB, Lolley RN. Cyclic guanosine monophosphate: elevation in degenerating photoreceptor cells of the C3H mouse retina. Science. 1974 Nov 1;186(4162):449-51. doi: 10.1126/science.186.4162.449. PMID 4369896
- [Background] Iribarne M, Masai I. Neurotoxicity of cGMP in the vertebrate retina: from the initial research on rd mutant mice to zebrafish genetic approaches. J Neurogenet. 2017 Sep;31(3):88-101. doi: 10.1080/01677063.2017.1358268. Epub 2017 Aug 16. PMID 28812418
- [Background] Vithana EN, Abu-Safieh L, Allen MJ, Carey A, Papaioannou M, Chakarova C, Al-Maghtheh M, Ebenezer ND, Willis C, Moore AT, Bird AC, Hunt DM, Bhattacharya SS. A human homolog of yeast pre-mRNA splicing gene, PRP31, underlies autosomal dominant retinitis pigmentosa on chromosome 19q13.4 (RP11). Mol Cell. 2001 Aug;8(2):375-81. doi: 10.1016/s1097-2765(01)00305-7. PMID 11545739
- [Background] Buskin A, Zhu L, Chichagova V, Basu B, Mozaffari-Jovin S, Dolan D, Droop A, Collin J, Bronstein R, Mehrotra S, Farkas M, Hilgen G, White K, Pan KT, Treumann A, Hallam D, Bialas K, Chung G, Mellough C, Ding Y, Krasnogor N, Przyborski S, Zwolinski S, Al-Aama J, Alharthi S, Xu Y, Wheway G, Szymanska K, McKibbin M, Inglehearn CF, Elliott DJ, Lindsay S, Ali RR, Steel DH, Armstrong L, Sernagor E, Urlaub H, Pierce E, Luhrmann R, Grellscheid SN, Johnson CA, Lako M. Disrupted alternative splicing for genes implicated in splicing and ciliogenesis causes PRPF31 retinitis pigmentosa. Nat Commun. 2018 Oct 12;9(1):4234. doi: 10.1038/s41467-018-06448-y. PMID 30315276
- [Background] Daiger SP, Sullivan LS, Bowne SJ. Genes and mutations causing retinitis pigmentosa. Clin Genet. 2013 Aug;84(2):132-41. doi: 10.1111/cge.12203. Epub 2013 Jun 19. PMID 23701314
- [Background] Yu DY, Cringle SJ, Su EN, Yu PK. Intraretinal oxygen levels before and after photoreceptor loss in the RCS rat. Invest Ophthalmol Vis Sci. 2000 Nov;41(12):3999-4006. PMID 11053305
- [Background] Usui S, Oveson BC, Lee SY, Jo YJ, Yoshida T, Miki A, Miki K, Iwase T, Lu L, Campochiaro PA. NADPH oxidase plays a central role in cone cell death in retinitis pigmentosa. J Neurochem. 2009 Aug;110(3):1028-37. doi: 10.1111/j.1471-4159.2009.06195.x. Epub 2009 May 30. PMID 19493169
- [Background] Shen J, Yang X, Dong A, Petters RM, Peng YW, Wong F, Campochiaro PA. Oxidative damage is a potential cause of cone cell death in retinitis pigmentosa. J Cell Physiol. 2005 Jun;203(3):457-64. doi: 10.1002/jcp.20346. PMID 15744744
- [Background] Komeima K, Usui S, Shen J, Rogers BS, Campochiaro PA. Blockade of neuronal nitric oxide synthase reduces cone cell death in a model of retinitis pigmentosa. Free Radic Biol Med. 2008 Sep 15;45(6):905-12. doi: 10.1016/j.freeradbiomed.2008.06.020. Epub 2008 Jun 28. PMID 18634866
- [Background] Komeima K, Rogers BS, Lu L, Campochiaro PA. Antioxidants reduce cone cell death in a model of retinitis pigmentosa. Proc Natl Acad Sci U S A. 2006 Jul 25;103(30):11300-5. doi: 10.1073/pnas.0604056103. Epub 2006 Jul 18. PMID 16849425
- [Background] Komeima K, Rogers BS, Campochiaro PA. Antioxidants slow photoreceptor cell death in mouse models of retinitis pigmentosa. J Cell Physiol. 2007 Dec;213(3):809-15. doi: 10.1002/jcp.21152. PMID 17520694
- [Background] Lee SY, Usui S, Zafar AB, Oveson BC, Jo YJ, Lu L, Masoudi S, Campochiaro PA. N-Acetylcysteine promotes long-term survival of cones in a model of retinitis pigmentosa. J Cell Physiol. 2011 Jul;226(7):1843-9. doi: 10.1002/jcp.22508. PMID 21506115
- [Background] Ait-Ali N, Fridlich R, Millet-Puel G, Clerin E, Delalande F, Jaillard C, Blond F, Perrocheau L, Reichman S, Byrne LC, Olivier-Bandini A, Bellalou J, Moyse E, Bouillaud F, Nicol X, Dalkara D, van Dorsselaer A, Sahel JA, Leveillard T. Rod-derived cone viability factor promotes cone survival by stimulating aerobic glycolysis. Cell. 2015 May 7;161(4):817-32. doi: 10.1016/j.cell.2015.03.023. PMID 25957687
- [Background] Petit L, Ma S, Cipi J, Cheng SY, Zieger M, Hay N, Punzo C. Aerobic Glycolysis Is Essential for Normal Rod Function and Controls Secondary Cone Death in Retinitis Pigmentosa. Cell Rep. 2018 May 29;23(9):2629-2642. doi: 10.1016/j.celrep.2018.04.111. PMID 29847794
- [Background] Campochiaro PA, Mir TA. The mechanism of cone cell death in Retinitis Pigmentosa. Prog Retin Eye Res. 2018 Jan;62:24-37. doi: 10.1016/j.preteyeres.2017.08.004. Epub 2017 Sep 27. PMID 28962928
- [Background] Aldini G, Altomare A, Baron G, Vistoli G, Carini M, Borsani L, Sergio F. N-Acetylcysteine as an antioxidant and disulphide breaking agent: the reasons why. Free Radic Res. 2018 Jul;52(7):751-762. doi: 10.1080/10715762.2018.1468564. Epub 2018 May 9. PMID 29742938
- [Background] Prescott LF, Park J, Ballantyne A, Adriaenssens P, Proudfoot AT. Treatment of paracetamol (acetaminophen) poisoning with N-acetylcysteine. Lancet. 1977 Aug 27;2(8035):432-4. doi: 10.1016/s0140-6736(77)90612-2. PMID 70646
- [Background] Smilkstein MJ, Knapp GL, Kulig KW, Rumack BH. Efficacy of oral N-acetylcysteine in the treatment of acetaminophen overdose. Analysis of the national multicenter study (1976 to 1985). N Engl J Med. 1988 Dec 15;319(24):1557-62. doi: 10.1056/NEJM198812153192401. PMID 3059186
- [Background] Decramer M, Rutten-van Molken M, Dekhuijzen PN, Troosters T, van Herwaarden C, Pellegrino R, van Schayck CP, Olivieri D, Del Donno M, De Backer W, Lankhorst I, Ardia A. Effects of N-acetylcysteine on outcomes in chronic obstructive pulmonary disease (Bronchitis Randomized on NAC Cost-Utility Study, BRONCUS): a randomised placebo-controlled trial. Lancet. 2005 Apr 30-May 6;365(9470):1552-60. doi: 10.1016/S0140-6736(05)66456-2. PMID 15866309
- [Background] Tse HN, Raiteri L, Wong KY, Yee KS, Ng LY, Wai KY, Loo CK, Chan MH. High-dose N-acetylcysteine in stable COPD: the 1-year, double-blind, randomized, placebo-controlled HIACE study. Chest. 2013 Jul;144(1):106-118. doi: 10.1378/chest.12-2357. PMID 23348146
- [Background] Zheng JP, Wen FQ, Bai CX, Wan HY, Kang J, Chen P, Yao WZ, Ma LJ, Li X, Raiteri L, Sardina M, Gao Y, Wang BS, Zhong NS; PANTHEON study group. Twice daily N-acetylcysteine 600 mg for exacerbations of chronic obstructive pulmonary disease (PANTHEON): a randomised, double-blind placebo-controlled trial. Lancet Respir Med. 2014 Mar;2(3):187-94. doi: 10.1016/S2213-2600(13)70286-8. Epub 2014 Jan 30. PMID 24621680
- [Background] Demedts M, Behr J, Buhl R, Costabel U, Dekhuijzen R, Jansen HM, MacNee W, Thomeer M, Wallaert B, Laurent F, Nicholson AG, Verbeken EK, Verschakelen J, Flower CD, Capron F, Petruzzelli S, De Vuyst P, van den Bosch JM, Rodriguez-Becerra E, Corvasce G, Lankhorst I, Sardina M, Montanari M; IFIGENIA Study Group. High-dose acetylcysteine in idiopathic pulmonary fibrosis. N Engl J Med. 2005 Nov 24;353(21):2229-42. doi: 10.1056/NEJMoa042976. PMID 16306520
- [Background] Idiopathic Pulmonary Fibrosis Clinical Research Network; Raghu G, Anstrom KJ, King TE Jr, Lasky JA, Martinez FJ. Prednisone, azathioprine, and N-acetylcysteine for pulmonary fibrosis. N Engl J Med. 2012 May 24;366(21):1968-77. doi: 10.1056/NEJMoa1113354. Epub 2012 May 20. PMID 22607134
- [Background] Idiopathic Pulmonary Fibrosis Clinical Research Network; Martinez FJ, de Andrade JA, Anstrom KJ, King TE Jr, Raghu G. Randomized trial of acetylcysteine in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2093-101. doi: 10.1056/NEJMoa1401739. Epub 2014 May 18. PMID 24836309
- [Background] Campochiaro PA, Iftikhar M, Hafiz G, Akhlaq A, Tsai G, Wehling D, Lu L, Wall GM, Singh MS, Kong X. Oral N-acetylcysteine improves cone function in retinitis pigmentosa patients in phase I trial. J Clin Invest. 2020 Mar 2;130(3):1527-1541. doi: 10.1172/JCI132990. PMID 31805012
- [Background] Usui S, Komeima K, Lee SY, Jo YJ, Ueno S, Rogers BS, Wu Z, Shen J, Lu L, Oveson BC, Rabinovitch PS, Campochiaro PA. Increased expression of catalase and superoxide dismutase 2 reduces cone cell death in retinitis pigmentosa. Mol Ther. 2009 May;17(5):778-86. doi: 10.1038/mt.2009.47. Epub 2009 Mar 17. PMID 19293779
- [Background] Xiong W, MacColl Garfinkel AE, Li Y, Benowitz LI, Cepko CL. NRF2 promotes neuronal survival in neurodegeneration and acute nerve damage. J Clin Invest. 2015 Apr;125(4):1433-45. doi: 10.1172/JCI79735. Epub 2015 Mar 23. PMID 25798616
- [Background] Kong X, Hafiz G, Wehling D, Akhlaq A, Campochiaro PA. Locus-Level Changes in Macular Sensitivity in Patients with Retinitis Pigmentosa Treated with Oral N-acetylcysteine. Am J Ophthalmol. 2021 Jan;221:105-114. doi: 10.1016/j.ajo.2020.08.002. Epub 2020 Aug 11. PMID 32795434
- [Background] Roberts PA, Gaffney EA, Whiteley JP, Luthert PJ, Foss AJE, Byrne HM. Predictive Mathematical Models for the Spread and Treatment of Hyperoxia-induced Photoreceptor Degeneration in Retinitis Pigmentosa. Invest Ophthalmol Vis Sci. 2018 Mar 1;59(3):1238-1249. doi: 10.1167/iovs.17-23177. PMID 29625444
- [Background] Cai CX, Locke KG, Ramachandran R, Birch DG, Hood DC. A comparison of progressive loss of the ellipsoid zone (EZ) band in autosomal dominant and x-linked retinitis pigmentosa. Invest Ophthalmol Vis Sci. 2014 Oct 23;55(11):7417-22. doi: 10.1167/iovs.14-15013. PMID 25342618
- [Background] Hariri AH, Zhang HY, Ho A, Francis P, Weleber RG, Birch DG, Ferris FL 3rd, Sadda SR; Trial of Oral Valproic Acid for Retinitis Pigmentosa Group. Quantification of Ellipsoid Zone Changes in Retinitis Pigmentosa Using en Face Spectral Domain-Optical Coherence Tomography. JAMA Ophthalmol. 2016 Jun 1;134(6):628-35. doi: 10.1001/jamaophthalmol.2016.0502. PMID 27031504
- [Background] Tee JJL, Yang Y, Kalitzeos A, Webster A, Bainbridge J, Michaelides M. Natural History Study of Retinal Structure, Progression, and Symmetry Using Ellipzoid Zone Metrics in RPGR-Associated Retinopathy. Am J Ophthalmol. 2019 Feb;198:111-123. doi: 10.1016/j.ajo.2018.10.003. Epub 2018 Oct 9. PMID 30312579
- [Background] FDA. E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials. https://www.fda.gov/regulatory-information/search-fda-guidance-documents/e9r1-statistical-principles-clinical-trials-addendum-estimands-and-sensitivity-analysis-clinical. 2019.
- [Background] Csaky K, Ferris F 3rd, Chew EY, Nair P, Cheetham JK, Duncan JL. Report From the NEI/FDA Endpoints Workshop on Age-Related Macular Degeneration and Inherited Retinal Diseases. Invest Ophthalmol Vis Sci. 2017 Jul 1;58(9):3456-3463. doi: 10.1167/iovs.17-22339. No abstract available. PMID 28702674
- [Background] O'Neal T, Luther E. Retinitis Pigmentosa. [Updated 2019 Apr 10]. In: Treasure Island (FL): StatPearls Publishing; 2019: https://www.ncbi.nlm.nih.gov/books/NBK519518/
- [Background] Sadda SR, Chakravarthy U, Birch DG, Staurenghi G, Henry EC, Brittain C. CLINICAL ENDPOINTS FOR THE STUDY OF GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2016 Oct;36(10):1806-22. doi: 10.1097/IAE.0000000000001283. PMID 27652913
- [Background] Linder B, Dill H, Hirmer A, Brocher J, Lee GP, Mathavan S, Bolz HJ, Winkler C, Laggerbauer B, Fischer U. Systemic splicing factor deficiency causes tissue-specific defects: a zebrafish model for retinitis pigmentosa. Hum Mol Genet. 2011 Jan 15;20(2):368-77. doi: 10.1093/hmg/ddq473. Epub 2010 Nov 3. PMID 21051334
- [Background] Birch DG, Cheng P, Duncan JL, Ayala AR, Maguire MG, Audo I, Cheetham JK, Durham TA, Fahim AT, Ferris FL 3rd, Heon E, Huckfeldt RM, Iannaccone A, Khan NW, Lad EM, Michaelides M, Pennesi ME, Stingl K, Vincent A, Weng CY; Foundation Fighting Blindness Consortium Investigator Group. The RUSH2A Study: Best-Corrected Visual Acuity, Full-Field Electroretinography Amplitudes, and Full-Field Stimulus Thresholds at Baseline. Transl Vis Sci Technol. 2020 Oct 8;9(11):9. doi: 10.1167/tvst.9.11.9. eCollection 2020 Oct. PMID 33133772
- [Background] Ramachandran R, X Cai C, Lee D, C Epstein B, Locke KG, G Birch D, C Hood D. Reliability of a Manual Procedure for Marking the EZ Endpoint Location in Patients with Retinitis Pigmentosa. Transl Vis Sci Technol. 2016 May 17;5(3):6. doi: 10.1167/tvst.5.3.6. eCollection 2016 May. PMID 27226930
- [Background] Sujirakul T, Lin MK, Duong J, Wei Y, Lopez-Pintado S, Tsang SH. Multimodal Imaging of Central Retinal Disease Progression in a 2-Year Mean Follow-up of Retinitis Pigmentosa. Am J Ophthalmol. 2015 Oct;160(4):786-98.e4. doi: 10.1016/j.ajo.2015.06.032. Epub 2015 Jul 9. PMID 26164827
- [Background] Iftikhar M, Kherani S, Kaur R, Lemus M, Nefalar A, Usmani B, Junaid N, Campochiaro PA, Scholl HPN, Shah SM. Progression of Retinitis Pigmentosa as Measured on Microperimetry: The PREP-1 Study. Ophthalmol Retina. 2018 May;2(5):502-507. doi: 10.1016/j.oret.2017.09.008. Epub 2017 Nov 9. PMID 31047333
- [Background] Tee JJL, Carroll J, Webster AR, Michaelides M. Quantitative Analysis of Retinal Structure Using Spectral-Domain Optical Coherence Tomography in RPGR-Associated Retinopathy. Am J Ophthalmol. 2017 Jun;178:18-26. doi: 10.1016/j.ajo.2017.03.012. Epub 2017 Mar 18. PMID 28322733
- [Background] Wilding GE, Chandrasekhar R, Hutson AD. A new linear model-based approach for inferences about the mean area under the curve. Stat Med. 2012 Dec 10;31(28):3563-78. doi: 10.1002/sim.5387. PMID 23175104
- [Background] Dawson JD. Sample size calculations based on slopes and other summary statistics. Biometrics. 1998 Mar;54(1):323-30. PMID 9544525
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Background] Little R, Rubin D. Statistical Analysis with Missing Data. Wiley; 2002
- [Background] SAS. SAS/STAT ® 14.1 User's Guide The MI Procedure. . 2015.
- [Background] Horton NJ, Lipsitz SR. Multiple imputation in practice: Comparison of software packages for regression models with missing variables. Am Stat. 2001;55(3):244-254.
- [Background] von Hippel PT. How to Impute Interactions, Squares and Other Transformed Variables. Sociol Methodol. 2009;39:265-291.
- [Background] Campion WM. Multiple Imputation for Nonresponse in Surveys - Rubin,Db. J Marketing Res. 1989;26(4):485-486
- [Background] Cabral T, Sengillo JD, Duong JK, Justus S, Boudreault K, Schuerch K, Belfort R Jr, Mahajan VB, Sparrow JR, Tsang SH. Retrospective Analysis of Structural Disease Progression in Retinitis Pigmentosa Utilizing Multimodal Imaging. Sci Rep. 2017 Sep 4;7(1):10347. doi: 10.1038/s41598-017-10473-0. PMID 28871101
- [Background] Hollander SA, Alsaleh N, Ruzhnikov M, Jensen K, Rosenthal DN, Stevenson DA, Manning M. Variable clinical course of identical twin neonates with Alstrom syndrome presenting coincidentally with dilated cardiomyopathy. Am J Med Genet A. 2017 Jun;173(6):1687-1689. doi: 10.1002/ajmg.a.38200. Epub 2017 Apr 13. PMID 28407410
- [Background] Alshamrani AA, Raddadi O, Schatz P, Lenzner S, Neuhaus C, Azzam E, Abdelkader E. Severe retinitis pigmentosa phenotype associated with novel CNGB1 variants. Am J Ophthalmol Case Rep. 2020 Jun 13;19:100780. doi: 10.1016/j.ajoc.2020.100780. eCollection 2020 Sep. PMID 32613137
- [Background] Iftikhar M, Usmani B, Sanyal A, Kherani S, Sodhi S, Bagheri S, Schonbach EM, Junaid N, Scholl HPN, Shah SMA. Progression of retinitis pigmentosa on multimodal imaging: The PREP-1 study. Clin Exp Ophthalmol. 2019 Jul;47(5):605-613. doi: 10.1111/ceo.13458. Epub 2019 Jan 2. PMID 30552737
- [Background] Birch DG, Locke KG, Wen Y, Locke KI, Hoffman DR, Hood DC. Spectral-domain optical coherence tomography measures of outer segment layer progression in patients with X-linked retinitis pigmentosa. JAMA Ophthalmol. 2013 Sep;131(9):1143-50. doi: 10.1001/jamaophthalmol.2013.4160. PMID 23828615
- [Background] Colombo L, Montesano G, Sala B, Patelli F, Maltese P, Abeshi A, Bertelli M, Rossetti L. Comparison of 5-year progression of retinitis pigmentosa involving the posterior pole among siblings by means of SD-OCT: a retrospective study. BMC Ophthalmol. 2018 Jun 26;18(1):153. doi: 10.1186/s12886-018-0817-z. PMID 29940899
- [Background] Takahashi VKL, Takiuti JT, Jauregui R, Lima LH, Tsang SH. Structural disease progression in PDE6-associated autosomal recessive retinitis pigmentosa. Ophthalmic Genet. 2018 Oct;39(5):610-614. doi: 10.1080/13816810.2018.1509354. Epub 2018 Aug 28. PMID 30153077
- [Background] Kim YN, Song JS, Oh SH, Kim YJ, Yoon YH, Seo EJ, Seol CA, Lee SM, Choi JM, Seo GH, Keum C, Lee BH, Lee JY. Clinical characteristics and disease progression of retinitis pigmentosa associated with PDE6B mutations in Korean patients. Sci Rep. 2020 Nov 11;10(1):19540. doi: 10.1038/s41598-020-75902-z. PMID 33177553
- [Background] Tee JJL, Yang Y, Kalitzeos A, Webster A, Bainbridge J, Weleber RG, Michaelides M. Characterization of Visual Function, Interocular Variability and Progression Using Static Perimetry-Derived Metrics in RPGR-Associated Retinopathy. Invest Ophthalmol Vis Sci. 2018 May 1;59(6):2422-2436. doi: 10.1167/iovs.17-23739. PMID 29847648
- [Background] Iftikhar M, Lemus M, Usmani B, Campochiaro PA, Sahel JA, Scholl HPN, Shah SMA. Classification of disease severity in retinitis pigmentosa. Br J Ophthalmol. 2019 Nov;103(11):1595-1599. doi: 10.1136/bjophthalmol-2018-313669. Epub 2019 Jan 31. PMID 30705041
- [Background] Permutt T. Sensitivity analysis for missing data in regulatory submissions. Stat Med. 2016 Jul 30;35(17):2876-9. doi: 10.1002/sim.6753. Epub 2015 Nov 15. PMID 26567763
- [Background] Kahan BC, Morris TP. Analysis of multicentre trials with continuous outcomes: when and how should we account for centre effects? Stat Med. 2013 Mar 30;32(7):1136-49. doi: 10.1002/sim.5667. Epub 2012 Oct 30. PMID 23112128
- [Background] Senn S. A note regarding 'random effects'. Stat Med. 2014 Jul 20;33(16):2876-7. doi: 10.1002/sim.5965. No abstract available. PMID 24898710
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Birch DG, Fish GE. Rod ERGs in retinitis pigmentosa and cone-rod degeneration. Invest Ophthalmol Vis Sci. 1987 Jan;28(1):140-50. PMID 3804644
- [Background] Birch DG, Wen Y, Locke K, Hood DC. Rod sensitivity, cone sensitivity, and photoreceptor layer thickness in retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2011 Sep 9;52(10):7141-7. doi: 10.1167/iovs.11-7509. PMID 21810977
- [Background] Dmitrienko A, D'Agostino R Sr. Traditional multiplicity adjustment methods in clinical trials. Stat Med. 2013 Dec 20;32(29):5172-218. doi: 10.1002/sim.5990. Epub 2013 Sep 30. PMID 24114861
- [Background] Papi A, Zheng J, Criner GJ, Fabbri LM, Calverley PMA. Impact of smoking status and concomitant medications on the effect of high-dose N-acetylcysteine on chronic obstructive pulmonary disease exacerbations: A post-hoc analysis of the PANTHEON study. Respir Med. 2019 Feb;147:37-43. doi: 10.1016/j.rmed.2018.12.014. Epub 2019 Jan 9. PMID 30704697
- [Background] Dmitrienko A, Muysers C, Fritsch A, Lipkovich I. General guidance on exploratory and confirmatory subgroup analysis in late-stage clinical trials. J Biopharm Stat. 2016;26(1):71-98. doi: 10.1080/10543406.2015.1092033. PMID 26366479
- [Background] Wang SJ, Hung HM. A regulatory perspective on essential considerations in design and analysis of subgroups when correctly classified. J Biopharm Stat. 2014;24(1):19-41. doi: 10.1080/10543406.2013.856022. PMID 24392976
- [Background] Dmitrienko A, D'Agostino RB Sr. Multiplicity Considerations in Clinical Trials. N Engl J Med. 2018 May 31;378(22):2115-2122. doi: 10.1056/NEJMra1709701. No abstract available. PMID 29847757
- [Background] Piantadosi S. Clinical trials : a methodologic perspective. 2005.
- [Background] Ying GS, Maguire MG, Glynn RJ, Rosner B. Tutorial on Biostatistics: Longitudinal Analysis of Correlated Continuous Eye Data. Ophthalmic Epidemiol. 2021 Feb;28(1):3-20. doi: 10.1080/09286586.2020.1786590. Epub 2020 Aug 2. PMID 32744149
- [Background] Zafarullah M, Li WQ, Sylvester J, Ahmad M. Molecular mechanisms of N-acetylcysteine actions. Cell Mol Life Sci. 2003 Jan;60(1):6-20. doi: 10.1007/s000180300001. PMID 12613655
- [Background] Echeverri-Ruiz N, Haynes T, Landers J, Woods J, Gemma MJ, Hughes M, Del Rio-Tsonis K. A biochemical basis for induction of retina regeneration by antioxidants. Dev Biol. 2018 Jan 15;433(2):394-403. doi: 10.1016/j.ydbio.2017.08.013. Epub 2017 Dec 25. PMID 29291983
- [Background] Oldham JM, Ma SF, Martinez FJ, Anstrom KJ, Raghu G, Schwartz DA, Valenzi E, Witt L, Lee C, Vij R, Huang Y, Strek ME, Noth I; IPFnet Investigators. TOLLIP, MUC5B, and the Response to N-Acetylcysteine among Individuals with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2015 Dec 15;192(12):1475-82. doi: 10.1164/rccm.201505-1010OC. PMID 26331942
- [Background] Moradi M, Mojtahedzadeh M, Mandegari A, Soltan-Sharifi MS, Najafi A, Khajavi MR, Hajibabayee M, Ghahremani MH. The role of glutathione-S-transferase polymorphisms on clinical outcome of ALI/ARDS patient treated with N-acetylcysteine. Respir Med. 2009 Mar;103(3):434-41. doi: 10.1016/j.rmed.2008.09.013. Epub 2008 Nov 7. PMID 18993042
- [Background] Zhang JQ, Zhang JQ, Liu H, Zhao ZH, Fang LZ, Liu L, Fu WP, Shu JK, Feng JG, Dai LM. Effect of N-acetylcysteine in COPD patients with different microsomal epoxide hydrolase genotypes. Int J Chron Obstruct Pulmon Dis. 2015 May 13;10:917-23. doi: 10.2147/COPD.S79710. eCollection 2015. PMID 25999707
- [Derived] Kong X, Ibukun F, Khan MJ, Hafiz G, Wehling D, Dreger K, Singh M, Birch D, Jaffe G, Naufal F, Traboulsi EI, Duncan J, Hufnagel R, Carroll J, Lu Y, Matsui R, Moulton LH, Hawkins B, Campochiaro PA; NAC Attack Study Investigative Group. Protocol for NAC Attack, a phase-3, multicenter randomized, parallel, double masked, placebo controlled trial evaluating the efficacy and safety of oral N-acetylcysteine (NAC) in patients with retinitis pigmentosa. medRxiv [Preprint]. 2025 Nov 6:2025.11.05.25339486. doi: 10.1101/2025.11.05.25339486. PMID 41282901
- See also: FDA. E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/e9r1-statistical-principles-clinical-trials-addendum-estimands-and-sensitivity-analysis-clinical
- See also: Description of retinitis pigmentosa — http://www.ncbi.nlm.nih.gov/books/NBK519518/
- See also: Sensitivity Analysis in Multiple Imputation for Missing Data: Sensitivity analysis for multiple interpolation of missing data — https://support.sas.com/resources/papers/proceedings14/SAS270-2014.pdf
- See also: DRCR. N. Anti-VEGF vs. Prompt Vitrectomy for VH From PDR - Full Text View - ClinicalTrials.gov — https://clinicaltrials.gov/ct2/show/NCT02858076
- See also: FDA. Guidance for Industry E9 Statistical Principles for Clinical Trials — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/e9-statistical-principles-clinical-trials